CLINICAL TRIAL: NCT07017816
Title: JACOB: Joint Administration of cDNA for TP53, checkpOint Inhibition and Boost/Hypofractionated Radiation. A Phase 0/1 Study in Children With Recurrent, Progressive or Refractory CNS Malignancies.
Brief Title: A Phase 0/1 Study of cDNA for TP53, Checkpoint Inhibition and Radiation in Children With Recurrent, Progressive or Refractory CNS Malignancies.
Acronym: JACOB
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Eugene Hwang, Professor of Pediatrics and Chief, Division of Oncology, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001415
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: CNS Malignancies; Medulloblastoma Recurrent; ATRT Recurrent; Pineoblastoma; Embryonal Neoplasm; Ependymoma Recurrent; High Grade Gliomas
MeSH Terms: conditions — Central Nervous System Neoplasms; Pinealoma; Neoplasms, Germ Cell and Embryonal | interventions — Immunotherapy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Patients with recurrent, progressive, or refractory CNS malignancies receiving SGT-53, Nivolumab, and radiation.
  Interventions: Drug: SGT-53; Radiation: hypofractionated radiotherapy with immunotherapy; Drug: Nivolumab

INTERVENTIONS:
Drug: SGT-53 — SGT-53 is a novel cationic liposome encapsulating a normal human wild type TP53 cDNA sequence in a plasmid backbone. The liposome is decorated on its surface with an anti- transferrin receptor (TfR) single chain antibody fragment (scFv) that is designed to target cancer cells through the binding of the TfRscFv to the transferrin receptor. This complex has been shown to efficiently and specifically deliver the TP53 complementary DNA (cDNA) to the tumor cells via receptor-mediated endocytosis of the cationic liposomal complex. Introduction of the TP53 cDNA sequence restores wild-type p53 (wtp53) function in the apoptotic pathway.
Radiation: hypofractionated radiotherapy with immunotherapy — Re-irradiation has rapidly grown into a primary consideration in the context of recurrent pediatric CNS malignancies. While not thought to be curative by itself, it has often resulted in temporary symptomatic improvement as well as occasional radiographic regression or stabilization, although as with any irradiation, may also cause some adverse events.
Drug: Nivolumab — Given the poor prognosis for children with recurrent CNS malignancies and the importance of p53 function in these tumors, we propose a pilot study of SGT-53 in combination with re-irradiation and checkpoint inhibition followed by maintenance therapy with SGT-53 in combination with nivolumab to evaluate the safety, feasibility and preliminary efficacy. SGT-53 will be added to a salvage regimen utilized in patients with recurrent tumors of re- irradiation and nivolumab followed by combination therapy with SGT-53 and nivolumab.

SUMMARY:
This clinical trial is studying a drug called SGT-53 along with radiation and another drug called Nivolumab. It's for children with brain tumors that have come back, gotten worse, or didn't get better with earlier treatments. The main questions it aims to answer are:

What is the right dose of SGT-53 that children can safely receive when it is used with radiation and Nivolumab? This dose will be used in the second phase of the trial.

What side effects are there of SGT-53 when it is used with radiation and Nivolumab?

How does SGT-53 move through the body when given with radiation and Nivolumab?

How much of the SGT-53 drug is found in the tumor tissue? This will be tested in a small group of patients?

Participants will:

For the first treatment cycle:

Get SGT-53 twice per week Get Nivolumab every 2 weeks Receive radiation therapy during week 2

For Cycles 2-6:

Get SGT-53 once per week during even cycles and twice per week during odd cycles Get Nivolumab every 2 weeks For Cycles 7+ Get both SGT-53 and Nivolumab every 2 weeks In the phase 0 part of the study, 4 participants will have genetic testing performed on their tumor tissue after receiving SGT-53. These samples will be compared to another sample taken from the skin.

ELIGIBILITY:
Inclusion Criteria:

* Tumor

  a. Patients must have a recurrent, progressive, or refractory CNS malignancy for which there are not known curative options.

  i. Medulloblastoma, ATRT, High grade gliomas, pineoblastomas, embryonal tumors NOS, CNS sarcomas, ependymomas, other high-grade malignancies that failed first line therapies.

ii. Patients should have received radiation for standard up-front therapy. iii. Patients must have received at least one line of standard of care treatment without limitation to the number of treatments received. b. Evidence of clinical and/or radiological progressive disease as defined by RAPNO criteria.

c. Patients with metastatic disease are eligible d. Patients must have available archival (formalin-fixed paraffin embedded) or fresh tumor tissue for correlative studies.

* Patient Characteristics a. The first 3 patients will be >7 years old to <22 years old i. Following initial successful treatment of the first 3 patients: Patients must be ≥3yrs and <22 years of age.

  b. Must have recovered from all surgical interventions prior to the start of the radiation and maintenance phases c. Patients must have a BSA of 0.6m2 or more to be enrolled. 3. Previous treatment
  1. Patients must have recovered from the acute effects of prior therapy. Adverse events resulting from prior surgical intervention will not be an ineligibility criterion.
  2. Chemotherapy: Patients must have received their last dose of known chemotherapy at least two (2) weeks prior to receipt of SGT-53.
  3. Biologic therapy: Patients must have received their last dose of biological agent >7 days prior to receipt of SGT-53.
  4. Radiation therapy: Patients must be deemed to be a reasonable candidate for hypofractionated irradiation from a clinical standard of care perspective.

  i. At least 3 months from craniospinal radiation therapy, ii. Other substantial bone marrow irradiation ≥6 weeks prior to enrollment, iii. Local palliative XRT (small volume) ≥2 weeks. iv. if progressive disease is documented by radiological evidence of disease in areas not previously radiated, no minimum time required.

  e. Corticosteroids: Patients who are receiving dexamethasone or other corticosteroids must be on a stable or decreasing dose for at least one (1) week prior to enrollment. There will be a maximum allowable steroid dose of 0.5mg/m2/day dexamethasone equivalents f. Growth factors: Patients must have received their last dose of any short acting growth factor at least one week prior to treatment, for long acting or pegylated growth factors, the last dose must be at least two (2) weeks prior to start of treatment.

  4. Neurologic Status

  a. Patients should be at their neurological baseline for a minimum of one week prior to enrollment.

  5. Performance Status

  a. Performance status (KarnofskyPS for >16yrs, or Lansky PS for <16yrs) assessed within two weeks must be >50.

  i. Patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for assessing the performance score.

  6. Organ Function - Patients must have normal organ and marrow function as defined below:
  1. Absolute neutrophil count >750/ul
  2. Platelets ≥75,000/ul
  3. Hemoglobin ≥8g/dL (may be supported with transfusion)
  4. Total bilirubin ≤1.5x ULN
  5. ALT/AST ≤3x ULN
  6. Serum albumin ≥2g/dL
  7. Normal cardiac function defined as ejection fraction within normal limits for age and gender
  8. a serum creatinine based on age/gender as below or a creatinine clearance or serum GFR ≥ 70ml/min/1.73m2: Serum Creatinine for age/sex Age Maximum Serum Creatinine (mg/dL) Male Female

     1. <2 years 0.6 0.6
     2. <6 years 0.8 0.8

     6-<10 years 1 1 10-<13 years 1.2 1.2 13- <16 years 1.5 1.4 > 16 years 1.7 1.4 The threshold creatinine values in this table were adapted from the Schwartz formula for estimating GFR (Schwartz et al. J. Peds 106:.522, 1985) utilizing child length and stature data published by the CDC.

     7. Pregnancy prevention- all patients of childbearing or child fathering potential must be willing to use an acceptable form of birth control while being treated on this study and at least 5 months after receiving the last study treatment.

     8. Pregnancy status: Female patients must not be pregnant or nursing. Female patients of reproductive potential must also have a negative serum pregnancy test at the time of enrollment.

     9. Informed Consent - Patient and/or guardian have the ability to understand and the willingness to sign a written informed consent document according to institutional guidelines.

     Exclusion Criteria:
* 1. Low-grade-glioma, craniopharyngioma, and other non-malignant CNS tumors are excluded.

  2. Patients with diagnosis of diffuse midline gliomas (DMGs) are excluded. 3. Patients with any clinically significant unrelated systemic illness (serious infection or significant cardiac, pulmonary, hepatic, or other organ dysfunction) that is likely to interfere with ability to tolerate study therapy or study procedure results.

  4. Patients with pre-existing cardiac dysfunction defined as baseline EF of less than 35% 5. Patients with pre-existing pulmonary fibrosis, interstitial lung disease, and clinically significant pulmonary lung disease.

  6. Patients who are receiving any other investigational drug therapy 7. Patients who in the opinion of the investigator cannot adhere to protocol requirements 8. Patients with history of autoimmune diseases that required treatment in the last 2 years are not eligible. Asymptomatic laboratory abnormalities (e.g. ANA, rheumatoid factor, altered thyroid function studies) will not render a patient ineligible in the absence of a diagnosis of an autoimmune disorder. Replacement therapy (e.g. thyroxine, insulin or physiologic corticosteroid replacement therapy) is not considered a form of systemic treatment.

  9. Patients who have received a live vaccine within 30 days of start of study treatment are not eligible.

  10. Patients with known HIV/AIDS or acute/chronic Hepatitis B or C are excluded.

  11. Patients who are prohibited from receiving radiation therapy (reached maximum lifetime dose) are not eligible.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Frequency and type of toxicity deemed at least probably related to SGT-53 | From enrollment to 3 years from end of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No